CLINICAL TRIAL: NCT06115083
Title: Long Term Effects of Pelvic Floor Re-education in Men With Chronic Pelvic Pain, Using Bio-feedback and Home Training - Subjective Outcomes in Correlation to Objective Measurements of the Lower Urinary Tract and Pelvic Floor
Brief Title: Effects of Pelvic Floor Training in Male Chronic Pelvic Pain, Correlation Between Subjective and Objective Outcomes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Stockholm (Other Government)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Lotta Renström Koskela, Principal Investigator, Region Stockholm
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: K 2023-4671
Record Dates: First submitted 2023-10-17; First posted 2023-11-02 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Chronic Pelvic Pain Syndrome; Chronic Prostatitis With Chronic Pelvic Pain Syndrome; Chronic Prostatitis; Pelvic Floor; Relaxation
Keywords: Chronic pelvic pain syndrome; Chronic prostatitis with chronic pelvic pain syndrome; Chronic prostatitis; Pelvic floor muscles; Urodynamics; Physiotherapy; Bio-feedback
MeSH Terms: conditions — Prostatitis

STUDY DESIGN:
Intervention Model Description: A randomized controlled single blinded clinical study with a study period of 12 months from inclusion until completion. The study subjects are then randomly assigned in a 1:1 ratio either to treatment or control group. After 6 months the study subjects in the control group are offered to be included in the intervention group.
Who Masked: Investigator
Masking Description: The interpreter of the urodynamic evaluations will be blinded regarding intervention/control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pelvic floor muscle re-education (Experimental): Intervention with pelvic floor re-education using bio-feedback and home training for 6 months, with a follow up visit after an additional period of 6 months
  Interventions: Other: Pelvic floor re-education using bio-feedback and home training
- Standard Care (No Intervention): No intervention during 6 months after inclusion. After the 6 month follow-up evaluation the study subjects are offered to participate in the interventional arm.

INTERVENTIONS:
Other: Pelvic floor re-education using bio-feedback and home training — Pelvic floor re-education using bio-feedback and home training
  Arms: Pelvic floor muscle re-education

SUMMARY:
The goal of this randomized controlled study is to establish the long-term effect of pelvic floor re-education using biofeedback and home training for men with chronic pelvic pain. The main questions it aims to answer are if pelvic floor re-education using bio-feedback and home training will give a long-lasting improvement in symptoms, assessed with a validated symptom score (the National Institute of Health - Chronic Prostatitis Symptom Index) and if an improvement in symptoms can be correlated to objective measurements of pelvic floor function. Participants will be asked to do pelvic floor exercises daily during six months with additional sessions of bio-feedback training. The control group will have no changes in their on-going treatment for their chronic pelvic pain and will be offered to enter the treatment group after six months.

DETAILED DESCRIPTION:
At baseline all included study subjects will fill in a validated symptom score, the National Institute of Health - Chronic Prostatitis Symptom Index (NIH-CPSI) and have an assessment of their pelvic floor muscles and undergo a urodynamic evaluation.

The intervention group will perform short daily session of pelvic floor muscle training at home during six months in combination with four bio-feedback sessions during the first months. The study subjects will receive an individual instruction based on the pelvic floor assessment from the baseline visit. The study subjects will report their training in a digital diary.

A reevaluation will be done at three, six and twelve months. At six and 12 months repeating the baseline tests. At three months a renewed assessment of muscle function and the NIH-CPSI questionnaire.

The control group will be instructed not to engage in any new treatment for their chronic pelvic pain during the study period. After the six months evaluation all participants in the control group will be offered to be enrolled in the treatment group, with the same set-up and follow-up as the treatment group.

ELIGIBILITY:
Inclusion Criteria:

* Men over the age of 18, residents in Sweden, diagnosed with Chronic Primary Pelvic Pain Syndrome (CPPPS) according to the International Statistical Classification of Diseases and Related Health Problems (ICD-10) (N41.1 (chronic prostatitis), N41.9 (Inflammatory disease of prostate, unspecified), N50.8F (Chronic Pelvic Pain Syndrome in men)

Exclusion Criteria:

* Cancer in the abdomen or pelvic organs (current or previous)
* Congenital anomalies affecting the pelvic region (Bladder exstrophy, Myelomeningocele etc.)
* Transsexual male, (i.e. at birth biologically female)
* Diseases affecting the nerve function to the pelvic and/or lower extremities, other disease or ongoing treatment that could have an impact on the outcome of the study.
* Incapability to participate in testing or follow training instructions due to mental incapacity, language difficulties etc.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in symptom score on the National Institute of Health-Chronic Prostatitis Symptom Index questionnaire | Measured 3, 6 and 12 months after inclusion
  Change in total score, range from 0-43 points. Higher score indicates worse symptoms.

SECONDARY OUTCOMES:
Change in sub score on the National Institute of Health-Chronic Prostatitis Symptom Index questionnaire | Measured 3, 6 and 12 months after inclusion
  Sub score according to the domains; pain 0-21, urological symptoms 0-10 points and quality of life impact 0-12 points. Higher score indicates worse symptoms in all three domains.
Changes in global voiding function using free flow non-invasive urodynamic testing | Measured 6 and 12 months after inclusion
  Changes in global voiding function using free flow non-invasive urodynamic testing with electromyogram.
  Global assessment where combined results from maximum urinary flow rate, voided volume, post voiding residual volume, pelvic floor activity during voiding and the shape of the curve are used to define types of voiding patterns.
  * Normal flow
  * Asymmetrical obstructive flow
  * Symmetrical low flow
  * Irregular curve, straining flow
  * Plateau low flow
  As described in the International Continence Society good urodynamic practices recommendations 2018 and Urodynamics (third edition) by P. Abrams.
Changes in global storing function of the bladder using invasive urodynamics, cystometry | Measured 6 and 12 months after inclusion
  Changes in global bladder function using invasive urodynamics with cystometry with electromyogram.
  Global assessment where combined results from sensory input, cystometric capacity, detrusor activity, compliance and pelvic floor activity are combined to define different patterns.
  * Normal cystometry
  * Abnormal sensory input
  * Detrusor activity
  * Abnormal compliance
  * Abnormal bladder capacity
  As described in the International Continence Society good urodynamic practices recommendations 2018 and Urodynamics (third edition) by P. Abrams.
Changes in global voiding function using invasive urodynamics, pressure-flow study | Measured 6 and 12 months after inclusion
  Changes in global voiding function using invasive urodynamics, pressure-flow study with electromyogram.
  Global assessment where combined results from detrusor contractility, urinary flow and pelvic floor activity are combined to define different patterns.
  * Normal flow
  * Under-active flow
  * Obstructed flow
  As described in the International Continence Society good urodynamic practices recommendations 2018 and Urodynamics (third edition) by P. Abrams.
Changes in urethral pressure using invasive urodynamics, urethral pressure profile | Measured 6 and 12 months after inclusion
  Changes in urethral pressure using invasive urodynamics, urethral pressure profile.
  * Maximum urethral pressure (cmH2O)
  * Maximum urethral closure pressure (cmH2O)
  As described in Urodynamics (third edition) by P. Abrams.
Changes in pelvic floor muscle assessment according to test specifics by Frawley et al 2021 and the modified Oxford Scale according to Laycock et al 2001. | Measured 3, 6 and 12 months after inclusion
  Pelvic floor muscle assessment according to test specifics by Frawley et al 2021
  1. Assessment of muscle tone
     - Decreased / normal / increased
  2. Assessment of voluntary contraction
     - No contraction / correct contraction / contraction only with help from other muscles / uncertain / straining
  3. Assessment of relaxation post contraction
     - Yes / partial or delayed / no
  4. Assessment of tenderness
     * Yes / No
     * If yes location is noted and severity of pain is graded according to numeric rating scale, 0-10, with higher value indicatinge more severe pain.
  Modified Oxford Scale for assessment of pelvic floor muscle power, graded from 0-5 with higer value indicating stronger power.
Correlation between subjective and objective measurements | Measured 3, 6 and 12 months after inclusion
  Correlation between subjective measurements using the National Institute of Health-Chronic Prostatitis Symptom Index questionnaire and objective findings on urodynamic testing and pelvic floor assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Lotta Renström Koskela, M.D, Principal Investigator — Karolinska University Hospital
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hallencreutz Grape H, Nordgren B, Renstrom Koskela L. Long-term effects of pelvic floor training in male chronic pelvic pain, correlation between subjective and objective outcomes: a study protocol for a randomised controlled trial. BMJ Open. 2024 Nov 4;14(11):e087620. doi: 10.1136/bmjopen-2024-087620. PMID 39496364